CLINICAL TRIAL: NCT02142764
Title: Preliminary Study for Selective Detection of the CD8+ Myelin Specific T Cell in the Blood of Multiple Sclerosis Patients (MS).
Brief Title: Preliminary Study for Selective Detection of the CD8+ Myelin Specific T Cell in the Blood of Multiple Sclerosis Patients
Acronym: IMMUNOSEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Merck Serono International SA (Industry); ADERA (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: CHUBX 2013/01
Record Dates: First submitted 2014-05-15; First posted 2014-05-20 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; CD8+ T-cells; Class I Major Histocompatibility Complex (MHC); pentamers
MeSH Terms: conditions — Multiple Sclerosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Multiple Sclerosis (Experimental): Human Leukocyte Antigen (HLA)-A2 patients whose Multiple Sclerosis has just been diagnosed
  Interventions: Biological: Blood samples
- Control (Other): HLA-A2 patients hospitalized in the neurology department who are not affected with a neuroimmunological disorder
  Interventions: Biological: Blood samples
- Multiple Sclerosis patients treated (Experimental): HLA-A2 Multiple Sclerosis patients treated by Natalizumab therapy
  Interventions: Biological: Blood samples

INTERVENTIONS:
Biological: Blood samples — The blood will be sampled in order to be tested in Immunology, twice, the day they sign their agreement and six months after in case of positive myelin pentamer test (at inclusion and 6 months after the inclusion).
  Arms: Multiple Sclerosis; Multiple Sclerosis patients treated
Biological: Blood samples — The blood will be sampled in order to be tested in Immunology, once, the day they sign their agreement (at the inclusion)
  Arms: Control

SUMMARY:
Most experts in the field consider Multiple Sclerosis as the main auto immune disease of the central nervous system. In spite of many works, the data in the literature concerning the antigens targeted by the CD8+ T-Cell response are still contradictory and insufficient.

DETAILED DESCRIPTION:
30 patients distributed in 3 groups of 10 patients with specific inclusion criteria will participate in this trial:

* 10 MS patients in early disease onset,
* 10 MS patients under Natalizumab treatment
* and control group of 10 patients with other neurological diseases.

The aim of this clinical trial is to detect the CD8+ myelin specific T-Cells in the blood of Multiple Sclerosis patients.

ELIGIBILITY:
Inclusion Criteria:

Group 1: HLA-A2 patients whose Multiple Sclerosis has just been diagnosed

* 18 year old and older patients,
* HLA-A2 Patients with Multiple Sclerosis or clinically isolated syndrome at high risk of being affected by Multiple Sclerosis (criteria of spatial scattering according to the 2010 or 2005 McDonald's criteria)
* Patients without treatment or treated with immunomodulating therapy
* Patients affiliated to health insurance coverage
* Information and comprehensive agreement signed by the patient and the investigator

Group 2: HLA-A2 patients hospitalized in the neurology department who are not affected with a neuroimmunological disorder

* 18 year old and older patients,
* HLA-A2 patients hospitalized in the neurology department
* Patient not affected by Multiple Sclerosis or a related inflammatory disorder
* Affiliated or profitable subject of a national insurance scheme
* Patients affiliated to health insurance coverage
* Information and comprehensive agreement signed by the patient and the investigator

Group 3: HLA-A2 Multiple Sclerosis patients treated by Natalizumab therapy

* 18 year old and older patients,
* HLA-A2 patients with relapsing remitting (RR) MS fulfilling McDonald 2005 or 2010 Multiple Sclerosis diagnostic criteria
* Patients treated by Natalizumab therapy for at least 3 months
* Patients affiliated to health insurance coverage
* Information and comprehensive agreement signed by the patient and the investigator

Exclusion Criteria:

Group 1 and 3:

* Patients undergoing immunosuppressive therapy at present or in the past except Natalizumab
* Pregnant women

Group 2:

* Patients undergoing immunosuppressive therapy at present or in the past
* Patients affected by Multiple Sclerosis or a related disorder
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Analysis of pentamers (> 0,1 % of the CD3 + CD8 + T-cells) will be statistically compared between the 3 groups of patients. | 6 months after the inclusion
  This analysis will enable us to detect CD8+ myelin specific T-cells in the blood of Multiple Sclerosis

SECONDARY OUTCOMES:
The results will be correlated with the patients clinical | 6 months after the inclusion
  Number of attacks relapses and evolution of the Expanded Disability Status Scale from the last 2 years
The results will be correlated with the patients MRI data | 6 months after the inclusion
  MRI activity (load lesions (≥ 9 lesions or not), gadolinium enhanced) from the last 2 years
Description of lymphocyte immunophenotyping and dosage of immunoglobulins in patients treated with Natalizumab | 6 months after the inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe OUALLET, MD, Principal Investigator — University Hospital Bordeaux, France
Locations (1):
- Service de Neurologie - Tripode - Hôpital Pellegrin, Bordeaux, Bordeaux, France